CLINICAL TRIAL: NCT07216963
Title: The Community Paramedic Response and Overdose Outreach With Supportive Medical-Legal Services (CROSSROADS) Study
Brief Title: The Community Paramedic Response and Overdose Outreach With Supportive Medical-Legal Services Study
Acronym: CROSSROADS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00118502; RM1DA064518 (NIH)
Record Dates: First submitted 2025-10-07; First posted 2025-10-15 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder; Overdose, Drug; Overdose; Substance Use (Drugs, Alcohol)
Keywords: Overdose; Community Paramedic; Medical-Legal Services; Criminal Legal System; Consolidated Framework for Implementation Research; Paramedical Personnel; Human Centered Design; Criminal Legal
MeSH Terms: conditions — Opioid-Related Disorders; Drug Overdose; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Paramedic Standard of Care (CP SOC) (Active Comparator): The community paramedic (CP) standard of care (SOC) has three basic components across all study sites. The core components of the CP SOC are that CPs: 1) are deployed via 911 as an opioid and/or stimulant overdose response; 2) provide Medications for Opioid Use Disorder (MOUD), harm reduction service referrals, and link patients to health and social programs as needed; and 3) provide long-term follow-up care in the field after initial contact.
  Interventions: Behavioral: Community Paramedic Standard of Care (CP SOC)
- CROSSROADS (Experimental): The community paramedic (CP) standard of care (SOC) has three basic components across the sites. The core components of the CP SOC are that CPs: 1) are deployed via 911 as an opioid and/or stimulant overdose response; 2) provide Medications for Opioid Use Disorder (MOUD), harm reduction service referrals, and link patients to health and social programs as needed; and 3) provide long-term follow-up care in the field after initial contact. The CROSSROADS intervention will utilize these SOC aspects and build in technology-supported medical-legal partnerships (MLP) via Docs for Health (D4H) that identifies and addresses health-harming legal needs (HHLN). While CP SOC may refer to services that address some HHLN, the key component of the CROSSROADS intervention is the direct identification and addressing of HHLN via D4H.
  Interventions: Behavioral: CROSSROADS

INTERVENTIONS:
Behavioral: Community Paramedic Standard of Care (CP SOC) — Participants randomized to CP SOC will receive 1) community paramedic standard of care after initial response to overdose; 2) Medications for Opioid Use Disorder (MOUD), harm reduction referrals, and linkages to health and social programs as needed; 3) long-term follow-up care with community paramedics in the field after initial contact.
  Arms: Community Paramedic Standard of Care (CP SOC)
Behavioral: CROSSROADS — The community paramedic (CP)standard of care (SOC) has three basic components across the sites. The core components of the CP SOC are that CPs: 1) are deployed via 911 as an opioid and/or stimulant overdose response; 2) provide Medications for Opioid Use Disorder (MOUD), harm reduction service referrals, and link patients to health and social programs as needed; and 3) provide long-term follow-up care in the field after initial contact. The CROSSROADS intervention will utilize these SOC aspects and build in technology-supported medical-legal partnerships (MLP) via Docs for Health (D4H) that identifies and addresses health-harming legal needs (HHLN). While CP SOC may refer to services that address some HHLN, the key component of the CROSSROADS intervention is the direct identification and addressing of HHLN via D4H.
  Arms: CROSSROADS

SUMMARY:
The goal of this clinical trial is to develop and test the CROSSROADS intervention. CROSSROADS is designed for people who have recently survived an opioid and/or stimulant-related non-fatal overdose and had contact with staff from a Community Paramedic (CP) program.

Participants will be randomly placed into one of two groups:

1) Standard of care from the CP program, or 2) CROSSROADS, which includes CP care plus a Medical-Legal Partnership (MLP). The MLP helps people with legal problems that can affect their health-- like issues with housing or public benefits.

Researchers will test if the CROSSROADS intervention reduces drug use and involvement with the criminal legal system.

People in the study will be followed for one year and asked to complete surveys at the beginning, and again at 1 month, 6 months, and 12 months.

DETAILED DESCRIPTION:
CROSSROADS is a Hybrid Type I Implementation Effectiveness Trial. The primary objective of the study is to examine how the CROSSROADS intervention, which incorporates a Medical-Legal Partnership (MLP) into community paramedic (CP) standard of care, addresses health-harming legal needs (HHLN) influencing adverse substance use outcomes and risk of CLS (Criminal Legal System) engagement.

The key component of the CROSSROADS intervention is that it directly identifies and addresses HHLN. The MLP utilized in this study is Docs for Health (D4H), a technology-supported mobile application MLP that utilizes a 'screen and intervene' approach.

The primary aim is to compare the CROSSROADS intervention versus standard of care (SOC) CP programs across four sites (Durham, NC; Miami, FL; Pittsburgh, PA; Portland, ME) on 1) frequency of opioid and stimulant use, and 2) CLS (police, incarceration, and probation/parole) involvement. Researchers will randomly assign 400 adults to the SOC CP program (n=200) or CROSSROADS (n=200). Follow-up will occur at 1, 6, and 12 months.

The focus of the study is to examine how Community paramedic programs addressing socio-structural-legal factors influence adverse substance use outcomes and risk of criminal legal engagement. The long-term goal is to assess how innovative non-carceral interventions can be best implemented to address adverse substance use outcomes and prevent CLS exposure.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older;
* Has interacted with a CP team (and, thus, experienced a non-fatal opioid and/or stimulant overdose) in the last 30 days;
* Has independent legal agency
* Able to independently provide informed consent; and
* Able to speak and understand English.

Exclusion Criteria:

- Active, severe, and untreated mental illness that would make providing consent impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of opioid and/or stimulant use | 12 months
  As measured by the number of days of use per month per participant.
Number of participants with opioid and/or stimulant use | 12 months
  As measured by Urine Drug Screen (UDS).
Number of participants with Criminal Legal System Involvement | 12 months
  Measured by the number of participants with criminal legal system involvement. Criminal legal system involvement includes all intercepts of the Sequential Intercept Model: police/arrest, jail, court, prison, and community supervision.

SECONDARY OUTCOMES:
Presence of Health Harming Legal Needs (HHLN) | 12 months
  Measured by the National Center for MLP HHLN Scale, which measures HHLN including income, education & employment, legal status, and personal stability. The scale "score" is the number of positive responses, indicating the number of identified legal needs a patient has on the screening tool.
Number of participants with risky substance use behaviors | 12 months
  Measured by the HIV Risk-taking Behavior Scale (HRBS). The HRBS provides three scores: a total score indicating level of HIV risk-taking behavior; a Drug Use Sub-total indicating level of risk due to drug taking practices; and a Sexual Behavior Sub-total indicating level of risk associated with unsafe sex. The higher the total score, the greater the risk the subject has of contracting and passing on HIV.
Risk of overdose as measured by the Opioid Overdose Risk Behavior Scale, version 2 (ORBS-2) | 12 months
  The total score on the ORBS-2 indicates the level of risk, with a higher score signifying a greater risk of overdose.
Number of participants who experienced a non-fatal overdose as measured by health record | 12 months
  Non-fatal overdoses measured by administrative/health records.
Number of participants who experienced a fatal overdose | 12 months
  Fatal overdoses are measured by administrative/health records.
Number of participants who utilized treatment services | 12 months
Number of participants who utilized overdose prevention services | 12 months
Number of participants who utilized harm reduction services | 12 months
Number of participants who utilized HHLN (Health Harming Legal Needs) ameliorative services | 12 months
  For example, eviction support, food stamps

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Brinkley-Rubinstein, PhD, Principal Investigator — Duke Health
Locations (4):
- United States (4):
  - University of Miami, Miami, Florida
  - Boston Medical Center, Boston, Massachusetts
  - Duke University, Durham, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No